CLINICAL TRIAL: NCT05920629
Title: Moderate Alcohol Consumption and Heart Function in Patients With a Recent Myocardial Infarction: a Multicentre Randomized Controlled Trial
Brief Title: Moderate Alcohol Consumption and Heart Function in Patients With a Recent Myocardial Infarction
Acronym: Moderate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baris Gencer (Other)
Collaborators: University of Bern (Other); Swiss National Science Foundation (Other)
Responsible Party: Sponsor-Investigator, Baris Gencer, Principal Investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-01838
Record Dates: First submitted 2023-02-14; First posted 2023-06-27 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Ethanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate alcohol consumption (No Intervention): 1 standard unit a day for 3 months
- Abstinence (Other): No alcohol beverages for 3 months
  Interventions: Behavioral: Alcohol consumption

INTERVENTIONS:
Behavioral: Alcohol consumption — After written consent, patients will enter a run-in period of 2 weeks where they will be asked not to drink any alcohol beverage. Patients with a successful run-in period will be randomized on a 1:1 basis stratified by baseline LVEF (<50% vs. ≥50%), sex and study site. 110 patients will be assigned to moderate alcohol consumption (1 standard unit a day), and 110 patients to abstinence (no alcohol beverages) for 3 months. We will perform a first echocardiography at randomization and a second at 3 months' follow-up.
  Arms: Abstinence

SUMMARY:
A total of 220 patients (110 per arm) who report moderate alcohol consumption between 4 and 28 standard units (1 standard unit = ~10 grams) per week in the 12 months prior to hospital admission will be planned for randomization, using a 1:1 ratio to pursue moderate alcohol consumption (1 standard unit per day for women and 2 standard units per day for men) or abstinence (except for one drink on predefined/agreed special occasions) for a total duration of 3 months. An echocardiography will be performed at baseline and 3 months to assess changes in systolic cardiac function (LVEF) for the primary endpoint. A core laboratory team blinded to assignment will perform data interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization for acute ST-elevation MI (STEMI) or non ST-elevation MI (NSTEMI) within 365 days prior to screening
* Men and women aged ≥18 years who are capable and willing to provide consent
* ECG ischemic changes, such as persistent or dynamic ST-segment deviation
* Evidence of positive high-sensitive troponin
* Confirmation of coronary heart disease aetiology by angiography
* Capacity to complete study visits with strict adherence to the protocol assignment
* Self-reported average alcohol consumption of between 4 and 28 standard units per week in the 12 months prior to the index hospitalization.

Exclusion Criteria:

* High alcohol consumption, defined as an average of >28 alcoholic standard units/week in the 12 months prior to the index hospitalization
* Alcohol use disorder (AUDIT score >20 at screening)
* History of alcohol or substance abuse
* Naïve to alcohol consumption
* Light alcohol consumption (<4 standard units by week)
* Prior severe heart failure (NYHA III-IV)
* Severe LV dysfunction at screening (<30%)
* History of gastric ulcer or gastro-intestinal bleeding
* Serious chronic liver disease or liver test elevation (> 3 times upper limit normal range)
* Personal history of any colon or liver cancer
* Any active malignancy (less than 5 years or ongoing treatment)
* Estimated glomerular filtration rate 15 ml/min/1.73m² or end-stage renal disease
* Any medication (investigator's discretion) making study participation impractical or precluding required follow-up
* History of organ transplant
* Participation in another trial testing intervention on similar CV outcomes (investigator's discretion)
* Any medical, geographic, or social factor making study participation impractical or precluding required follow-up.
* Pregnant, breastfeeding or planning to become pregnant within 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Cardiac function | 3 months
  Measurement of change in left ventricular ejection fraction between baseline visit and 3-month visit

CONTACTS AND LOCATIONS:
Overall Officials: Baris Gencer, MD, Principal Investigator — CHUV
Locations (3):
- Switzerland (3):
  - Centre hospitalier universitaire vaudois, Lausanne, Canton of Vaud
  - Inselspital, Bern
  - Hôpitaux Universitaires de Genève, Geneva